CLINICAL TRIAL: NCT06011473
Title: Continuous Glucose Monitoring for Colorectal Cancer
Acronym: CGM-CRC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NKBBN/780/2022
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Continuous Glucose Monitoring; Colorectal Cancer
Keywords: cgm; Colorectal Cancer; continuous glucose monitoring
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Study subjects submitted to the General Surgery Clinic for colorectal surgery. On admission day, patients will have a CGM sensor placed on the outer part of the upper arm. Patients will undergo standard surgical procedures and perioperative care. Glycemia will be continuously monitored for 10 days. The CGM sensor will be taken off during visit in Outpatient Clinic.
  Interventions: Device: CGM (FreeStyle Libre 3)

INTERVENTIONS:
Device: CGM (FreeStyle Libre 3) — FreeStyle Libre 3 system consists of a sensor that measures interstitial glycemia every minute and a dedicated application on mobile phone. Measurements are transmitted via Bluetooth to a mobile phone, that collects the data in the mobile application. Moreover, the study subject's application is connected to the doctor's application which allows remote real-time glycemia monitoring on another device.
  Other Name: continuous glucose monitoring, CGM, FreeStyle Libre 3

SUMMARY:
Hyperglycemia commonly occurs during surgery due to a reaction to metabolic stress and trauma. It has been shown that improper glycemia control leads to impaired wound healing and a higher risk of other postoperative complications.

The primary aim of our project is to assess the feasibility of the use of continuous glucose monitoring in measuring blood glucose levels in patients undergoing colorectal cancer surgery. The secondary aim is to analyze changes in perioperative blood glucose levels to understand the effects of stress and intraoperative interventions on the blood glucose level. The tertiary goal is to assess the predictive value of hyperglycemia for surgical site infection.

DETAILED DESCRIPTION:
Hyperglycemia commonly occurs during surgery due to a reaction to metabolic stress and trauma. It has been shown that improper glycemia control leads to impaired wound healing and a higher risk of other postoperative complications. However, glucose levels measured in patients before surgery are taken infrequently, and there remains controversy regarding optimal management. Usually, a blood glucose meter is used to measure non-fasted blood glucose concentrations, and a single-point measurement can easily misrepresent the actual glycemic control. Continuous glucose monitoring allows for a minimally invasive real-time remote glycemia control and is providing insights into glucose regulation in patients, demonstrating significant periods of clinically silent hypoglycemia and hyperglycemia.

The primary aim of our project is to assess the feasibility of the use of CGM in measuring blood glucose levels in patients undergoing colorectal cancer surgery. The secondary aim is to analyze changes in perioperative blood glucose levels to understand the effects of stress and intraoperative interventions on the blood glucose level. The tertiary goal is to assess the predictive value of hyperglycemia for surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* confirmed colorectal cancer qualified for surgery

Exclusion Criteria:

* patients who will be unable or will refuse to express informed concern
* pregnant women
* people undergoing dialysis treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-27 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
feasibility of CGM system | 10 days
  measured as the drop-out rate caused by non-adherence of both patients and medical staff due to system detaching, problems with the receiving device (low battery. distance beyond Bluetooth communication range) etc.

SECONDARY OUTCOMES:
perioperative glycemia | 10 days
  number of hyperglycemia episodes impact of stress and intraoperative interventions on the blood glucose level
SSI rate | 30 days
  Surgical Site Infection according to Centre for Disease Control criteria:
  Infection occurring within the first 30 post-operative days with at least one of the following:
  Purulent drainage from the incision Organisms isolated from an aseptically obtained culture of fluid or tissue from the incision
  Incision is deliberately opened by a surgeon AND at least one of the following signs/symptoms of infection:
  Pain or tenderness Localized swelling Redness Heat Diagnosis of SSI by the surgeon or attending physician

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Antoszewska, MD, Principal Investigator — MUG Division of Dermatology, Venereology and Allergology; Piotr Spychalski, MD, PhD, Principal Investigator — MUG Division of General Surgery; Jarosław Kobiela, Prof., Principal Investigator — MUG Division of General Surgery
Locations (1):
- UCC Division of Oncological, Transplant and General Surgery, Gdansk, Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McConnell YJ, Johnson PM, Porter GA. Surgical site infections following colorectal surgery in patients with diabetes: association with postoperative hyperglycemia. J Gastrointest Surg. 2009 Mar;13(3):508-15. doi: 10.1007/s11605-008-0734-1. Epub 2008 Nov 11. PMID 19002535